CLINICAL TRIAL: NCT06311071
Title: The Utility of Coronary Artery Calcium Score for the Prediction of Coronary Artery Disease in Patients With Cardiac Symptoms; a Diagnostic Study
Brief Title: The Predictive Value of Coronary Artery Calcium Score
Status: Completed | Type: Observational
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Other Study IDs: IR.SUMS.MED.REC.1401.200
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; coronary calcium score; cardiovascular risk score
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 365 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient group: patient suspected to have coronary artery disease in noninvasive tests
  Interventions: Diagnostic Test: calcium score; Diagnostic Test: Invasive coronary angiography

INTERVENTIONS:
Diagnostic Test: calcium score — Calcium score of coronaries obtained fro coronary CT angiography
  Other Names: CAC score
Diagnostic Test: Invasive coronary angiography — Invasive coronary angiography from radial artery with contrast injection

SUMMARY:
In this analytical prospective study 498 patients over 40 years with any cardiovascular symptoms and without pre-established coronary artery disease ( CAD) were enrolled. Patients underwent CT scans to measure coronary artery calcium score (CACS), and total calcium scores were recorded. Then, conventional coronary angiography was performed for all the participants as the gold standard for diagnosing CAD (defined as at least one stenotic coronary artery with ≥ 50%). Framingham risk score (FRS) was also estimated for all the patients

DETAILED DESCRIPTION:
In this prospective study 498 patient who referred to cardiology clinic with any cardiac symptoms and positive noninvasive tests without preestablished coronary artery disease ( CAD), were enrolled. All the patients underwent coronary artery calcium score (CACS) testing, and total calcium scores were recorded. A calcium score of zero was considered as having very low risk for CAD. A score of 1 to 99 was defined as having low risk, 101 to 299 as having intermediate risk, and 400 or more as having high risk for CAD. Then, invasive (conventional) coronary angiography by radial access, as the gold standard for the diagnosis of CAD, was performed for all of the involved participants.

Coronary artery stenosis equal to or more than 50% was considered as a significant narrowing [25]. Patients with at least one diseased coronary artery with a significant narrowing were considered to have CAD. Minor branches were considered only if their main supplying branch was not diseased. A group of expert interventional cardiologists performed and reported coronary angiographies. The study was single-blind; cardiologists were unaware of the results of CAC scores when performing conventional coronary angiographies

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years, having cardiovascular symptoms (including chest pain, dyspnea on exertion, etc.), and positive primary non-invasive tests, such as myocardial perfusion imaging (MPI) or exercise tolerance test (ETT)

Exclusion Criteria:

* Previously diagnosed coronary artery disease
* Cerebrovascular accident (CVA)
* Peripheral artery disease
* Pregnancy
* Medical instability
* Hypersensitivity to contrast materials
* Having atrial fibrillation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with any cardiac symptoms with positive noninvasive tests referred to cardiology clinic with positive non invasive tests like exercise test or echocardiography or perfusion cardiac scan
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
coronary artery disease | 1 year
  stenosis more than 50% in selective coronary angiography
coronary calcium score | 1 year
  calcium score obtained from coronary CT angiography, 0 no risk, 0-100 low risk, more than 100 high risk

SECONDARY OUTCOMES:
cardiovascular risk score | 1 year
  cardiovascular risk score obtained from Framingham risk score, low risk if less than 10%, moderate risk 10-20% and high risk if more than 20%

CONTACTS AND LOCATIONS:
Locations (1):
- Javad Kojuri, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: No
The data is available in registry and will be available on rational request